CLINICAL TRIAL: NCT06155487
Title: A Randomized, Double-blind, Placebo-controlled, Single and Multiple Ascending Dose, Phase 1 Clinical Trial to Evaluate Pharmacokinetics, Pharmacodynamics, Safety and Tolerability After Oral Administration of AJH-2947 in Healthy Korean or Caucasian Male Subjects
Brief Title: A Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics After Oral Administration of AJH-2947 in Healthy Korean and/or Caucasian Adult Male Subjects
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: JMackem Co., Ltd (Industry)
Collaborators: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AJH-2947_101
Record Dates: First submitted 2023-11-16; First posted 2023-12-04 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Neuropathic Pain; Diabetic Neuropathies; Post Herpetic Neuralgia
Keywords: Neuropathic Pain; TRPV1 antagonist; Phase 1
MeSH Terms: conditions — Neuralgia; Diabetic Neuropathies; Neuralgia, Postherpetic | interventions — Sagittal Abdominal Diameter; mycophenolic adenine dinucleotide

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, placebo-controlled, single and multiple ascending dose
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- (Part A) Single dose group 1 (Experimental): Oral dose of AJH-2947/placebo 100 mg, Korean Only*
  Interventions: Drug: AJH-2947 100 mg (SAD); Drug: Placebo
- (Part A) Single dose group 2 (Experimental): Oral dose of AJH-2947/placebo 200 mg, Korean and Caucasian
  Interventions: Drug: AJH-2947 200 mg (SAD); Drug: Placebo
- (Part A) Single dose group 3 (Experimental): Oral dose of AJH-2947/placebo 300 mg, Korean and Caucasian
  Interventions: Drug: AJH-2947 300 mg (SAD); Drug: Placebo
- (Part A) Single dose group 4 (Experimental): Oral dose of AJH-2947/placebo 400 mg, Korean and Caucasian
  Interventions: Drug: AJH-2947 400 mg (SAD); Drug: Placebo
- (Part A) Single dose group 5 (Experimental): Oral dose of AJH-2947/placebo 600 mg, Korean and Caucasian
  Interventions: Drug: AJH-2947 600 mg (SAD); Drug: Placebo
- (Part A) Single dose group 6 (Experimental): Oral dose of AJH-2947/placebo 800 mg, Korean and Caucasian
  Interventions: Drug: AJH-2947 800 mg (SAD); Drug: Placebo
- (Part B) Multiple dose group 1 (Experimental): Oral dose of AJH-2947/placebo 200 mg, Korean and Caucasian
  Interventions: Drug: AJH-2947 200 mg (MAD); Drug: Placebo
- (Part B) Multiple dose group 2 (Experimental): Oral dose of AJH-2947/placebo 400 mg, Korean and Caucasian
  Interventions: Drug: AJH-2947 400 mg (MAD); Drug: Placebo
- (Part B) Multiple dose group 3 (Experimental): Oral dose of AJH-2947/placebo 600 mg, Korean and Caucasian
  Interventions: Drug: AJH-2947 600 mg (MAD); Drug: Placebo

INTERVENTIONS:
Drug: AJH-2947 100 mg (SAD) — Oral Tablet, Single dose of AJH-2947 100 mg
  Arms: (Part A) Single dose group 1
Drug: Placebo — Oral Tablet, Single dose of Placebo 100 mg
  Arms: (Part A) Single dose group 1
Drug: AJH-2947 200 mg (SAD) — Oral Tablet, Single dose of AJH-2947 200 mg
  Arms: (Part A) Single dose group 2
Drug: Placebo — Oral Tablet, Single dose of Placebo 200 mg
  Arms: (Part A) Single dose group 2
Drug: AJH-2947 300 mg (SAD) — Oral Tablet, Single dose of AJH-2947 300 mg
  Arms: (Part A) Single dose group 3
Drug: Placebo — Oral Tablet, Single dose of Placebo 300 mg
  Arms: (Part A) Single dose group 3
Drug: AJH-2947 400 mg (SAD) — Oral Tablet, Single dose of AJH-2947 400 mg
  Arms: (Part A) Single dose group 4
Drug: Placebo — Oral Tablet, Single dose of Placebo 400 mg
  Arms: (Part A) Single dose group 4
Drug: AJH-2947 600 mg (SAD) — Oral Tablet, Single dose of AJH-2947 600 mg
  Arms: (Part A) Single dose group 5
Drug: Placebo — Oral Tablet,Single dose of Placebo 600 mg
  Arms: (Part A) Single dose group 5
Drug: AJH-2947 800 mg (SAD) — Oral Tablet, Single dose of AJH-2947 800 mg
  Arms: (Part A) Single dose group 6
Drug: Placebo — Oral Tablet, Single dose of Placebo 800 mg
  Arms: (Part A) Single dose group 6
Drug: AJH-2947 200 mg (MAD) — Oral Tablet, Multiple (once daily for 7days) oral dose of AJH-2947 200 mg
  Arms: (Part B) Multiple dose group 1
Drug: Placebo — Oral Tablet, Multiple (once daily for 7days) oral dose of Placebo 200 mg
  Arms: (Part B) Multiple dose group 1
Drug: AJH-2947 400 mg (MAD) — Oral Tablet,Multiple (once daily for 7days) oral dose of AJH-2947 400 mg
  Arms: (Part B) Multiple dose group 2
Drug: Placebo — Oral Tablet, Multiple (once daily for 7days) oral dose of Placebo 400 mg
  Arms: (Part B) Multiple dose group 2
Drug: AJH-2947 600 mg (MAD) — Oral Tablet, Multiple (once daily for 7days) oral dose of AJH-2947 600 mg
  Arms: (Part B) Multiple dose group 3
Drug: Placebo — Oral Tablet, Multiple (once daily for 7days) oral dose of Placebo 600 mg
  Arms: (Part B) Multiple dose group 3

SUMMARY:
Preliminary evaluate of pharmacokinetics, pharmacodynamics, safety and tolerability after oral administration of AJH-2947 in healthy Korean or Caucasian male subjects

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Korean or Caucasian adult males aged 19 to 55 years old, based on the date of written consent

   *Caucasian subjects = Individuals born in Europe, have resided in countries outside Europe for less than 10 years, and whose parents and grandparents are all of European descent.
2. Individuals with a body weight between 50.0 kg and 90.0 kg and a body mass index (BMI) ranging from 18.5 kg/m2 to less than 30.0 kg/m2

   - BMI (kg/m2) = weight (kg) / {height (m)}2
3. Individuals who agree to stay in the CTC ward until discharge and consent to the use of sunscreen until the end of the clinical trial (PSV)
4. Individuals who have heard a detailed explanation of the trial, fully understand it, voluntarily decide to participate, and provide written consent before the screening examination
5. Individuals deemed suitable by the investigator based on medical history, vital signs, 12-lead electrocardiogram (ECG), physical examination, and clinical laboratory tests performed during the screening.

Exclusion Criteria:

1. Individuals with clinically significant diseases or a history of diseases related to the liver, kidney, nervous system, immune system, respiratory system, digestive system, endocrine system, blood/tumors, cardiovascular system, urinary system, mental disorders, etc.
2. In the multiple-dose trial, individuals with skin lesions, tattoos on both forearms or show hypersensitivity or allergic reactions to capsaicin cream who may affect the pharmacodynamic evaluation of the investigational product.
3. Individuals with gastrointestinal diseases (such as gastrointestinal ulcers, gastritis, gastric spasm, gastroesophageal reflux disease, and Crohn's disease) or a history of surgery that may affect the safety and pharmacokinetic evaluation of the investigational product (excluding simple appendectomy and hernia repair)
4. Individuals with a medical history of hypersensitivity reactions to the main active ingredient or components of the investigational product or to drugs in the same class as the main active ingredient
5. Individuals with positive results for hepatitis B (HBV) test, hepatitis C (HCV) test, syphilis (RPR) test, or HIV test conducted during screening
6. Individuals who exhibited systolic blood pressure < 80 mmHg or ≥ 140 mmHg or diastolic blood pressure < 45 mmHg or ≥ 90 mmHg during vital sign measurements in the supine position after a rest period of at least three minutes
7. Individuals with a history of drug abuse or who tested positive for drug abuse in the urine drug screening test
8. Individuals who have taken prescription drugs or traditional herbal medicine within 2 weeks before the scheduled first dose of the investigational product or have taken any over-the-counter medicines, health-functional foods, or vitamin supplements within 1 week, or are expected to take them
9. Individuals who have participated in another clinical trial (including bioequivalence studies) within 6 months before the scheduled first dose of the investigational product
10. Individuals who donated blood within 2 months or donated blood components within 1 month, or received a blood transfusion within 1 month before the scheduled first dose of the investigational product
11. Individuals who have consumed excessive caffeine (> 5 units/day) or cannot abstain from consuming caffeine/caffeine-containing foods (such as coffee, tea, carbonated beverages, coffee-flavored milk, energy drinks, etc.) from 3 days before the expected first dose until the end of the clinical trial (PSV)
12. Individuals who engage in persistent alcohol consumption (> 21 units/week, 1 unit = 10 g of pure alcohol) or cannot abstain from alcohol consumption from 3 days before the expected first dose of the investigational product until the end of the clinical trial (PSV) (1 glass (250 mL) of beer (5%) = 10 g, 1 glass (50 mL) of soju (20%) = 8 g, 1 glass (125 mL) of wine (12%) = 12 g)
13. Individuals who have smoked more than 10 cigarettes/day within the last 3 months before the scheduled first dose of the investigational product or cannot quit smoking from the screening day until the end of the clinical trial (PSV)
14. Individuals who cannot refrain from consuming grapefruit-containing foods from 3 days before the expected first dose of the investigational product until the end of the clinical trial (PSV)
15. Individuals who have a pregnancy planning during the entire clinical trial and up to 90 days after the last administration of the investigational product or do not agree to use one or more medically acceptable contraceptive methods. The medically acceptable contraceptive methods are as follows:

    ① Use of an intrauterine device with a proven failure rate by the spouse (or partner)

    ② Concurrent use of barrier contraception (male or female) and oral contraceptive pills

    ③ Self or partner's surgical sterilization (vasectomy, salpingectomy / tubal ligation, hysterectomy)
16. Individuals deemed ineligible for participation in the clinical trial by the investigator based on other reasons, including results of clinical laboratory tests

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2023-12-05 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Part A (SAD): Plasma concentrations of AJH-2947 | Day 1 to Day 5
  To characterize the plasma concentration of AJH-2947 after single oral dosing in healthy Korean and Caucasian male participants.
Part A (SAD): Urine concentrations of AJH-2947 | Day 1 to Day 4
  To characterize the urine concentration of AJH-2947 after single oral dosing in healthy Korean and Caucasian male participants.
Part A (SAD): Maximum observed concentration [Cmax] | Day 1 to Day 5
  To characterize the Cmax of AJH-2947 after single oral dosing in healthy Korean and Caucasian male participants
Part A (SAD): Area under concentration curve from time 0 to the last quantifiable concentration [AUClast] | Day 1 to Day 5
  To characterize the AUClast of AJH-2947 after single oral dosing in healthy Korean and Caucasian male participants.
Part A (SAD): Time to reach peak or maximum observed concentration [Tmax] | Day 1 to Day 5
  To characterize the Tmax of AJH-2947 after single oral dosing in healthy Korean and Caucasian male participants.
Part B (MAD): Plasma concentrations of AJH-2947 | Day 1 to Day 18
  To characterize the plasma concentration of AJH-2947 following oral administration of multiple ascending doses in healthy Korean and Caucasian male participants.
Part B (MAD): Maximum observed concentration [Cmax] | Day 1 to Day 18
  To characterize the Cmax of AJH-2947 following oral administration of multiple ascending doses in healthy Korean and Caucasian male participants.
Part B (MAD): The partial area from dosing time to dosing time plus dosing interval [AUCτ] | Day 1 to Day 18
  To characterize the AUCτ of AJH-2947 following oral administration of multiple ascending doses in healthy Korean and Caucasian male participants.
Part B (MAD): Time of maximum observed concentration [Tmax] | Day 1 to Day 18
  To characterize the Tmax of AJH-2947 following oral administration of multiple ascending doses in healthy Korean and Caucasian male participants.
Part B (MAD): Maximum observed concentration occurring at time Tmax,ss [Cmax,ss] | Day 1 to Day 18
  To characterize the Cmax,ss of AJH-2947 following oral administration of multiple ascending doses in healthy Korean and Caucasian male participants.
Part B (MAD): At steady state, the partial area from dosing time to dosing time plus dosing interval [AUCτ,ss] | Day 1 to Day 18
  To characterize the AUCτ,ss of AJH-2947 following oral administration of multiple ascending doses in healthy Korean and Caucasian male participants.
Part B (MAD): Heat pain Threshold (The temperature at which the subject first perceives pain, ℃) | Predose, Day 1, Day 7, and Day 8
  Heat pain Threshold is determined by gradually increased the temperature of the thermal probe on non-sensitized and casaicin-sensitized skin starting from 30 ℃ as the baseline using Thermal NeuroSensory Analyzer. (The cutoff limit is set at 50°C)
Part B (MAD): Heat pain tolerance (The Maximum temperature that the subject can tolerate, ℃) | Predose, Day 1, Day 7, and Day 8
  Heat pain tolerance is determined by gradually increased the temperature of the thermal probe on non-sensitized and casaicin-sensitized skin starting from 30 ℃ as the baseline using Thermal NeuroSensory Analyzer. (The cutoff limit is set at 50°C)

SECONDARY OUTCOMES:
Part A (SAD): Number of participants with adverse events (AE) | Day -1, Day 1 to day 12 (last visit)
  To assess the safety and tolerability of AJH-2947 following oral administration of single ascending doses in healthy Korean and Caucasian male participants.
Part A (SAD): Number of participants with serious adverse events (SAE) | Day -1, Day 1 to day 18 (last visit)
  To assess the safety and tolerability of AJH-2947 following oral administration of multiple ascending doses in healthy Korean and Caucasian male participants.
Part B (MAD): Number of participants with AE | Day -1, Day 1 to day 18 (last visit)
  To assess the safety and tolerability of AJH-2947 following oral administration of multiple ascending doses in healthy Korean and Caucasian male participants.
Part B (MAD): Number of participants with SAE | Day -1, Day 1 to day 18 (last visit)
  To assess the safety and tolerability of AJH-2947 following oral administration of multiple ascending doses in healthy Korean and Caucasian male participants.

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Hwan Lee, MD. Ph.D, Principal Investigator — Seoul National University Clinical Trials Center
Locations (1):
- Seoul National University Hospital, Seoul, South Korea